CLINICAL TRIAL: NCT06399419
Title: An Open-Label, Phase I, Dose-Finding Study of CBM588 in Combination With Nivolumab/Ipilimumab for Patients With Advanced Stage Renal Cell Carcinoma
Brief Title: CBM588 Capsules in Combination With Nivolumab and Ipilimumab for the Treatment of Advanced Stage Kidney Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Osel, Inc. (Industry)
Collaborators: City of Hope Medical Center (Other); Miyarisan Pharmaceuticals, Co., Ltd. (Unknown); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23554; NCI-2024-03079 (Registry Identifier: Registry Identifier: CTRP (Clinical Trial Reporting Program)); 23554 (Other: City of Hope Comprehensive Cancer Center); P30CA033572 (NIH); NCT06414642 (obsolete NCT alias)
Record Dates: First submitted 2024-05-01; First posted 2024-05-03 (Actual); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Advanced Clear Cell Renal Cell Carcinoma; Advanced Renal Cell Carcinoma; Advanced Sarcomatoid Renal Cell Carcinoma; Metastatic Clear Cell Renal Cell Carcinoma; Metastatic Renal Cell Carcinoma; Metastatic Sarcomatoid Renal Cell Carcinoma; Stage III Renal Cell Cancer AJCC v8; Stage IV Renal Cell Cancer AJCC v8
MeSH Terms: conditions — Clear-cell metastatic renal cell carcinoma; Carcinoma, Renal Cell | interventions — Specimen Handling; Ipilimumab; CTLA-4 Antigen; Magnetic Resonance Spectroscopy; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (CBM588 capsules, nivolumab, ipilimumab) (Experimental): Patients receive CBM588 PO BID on days 1-21, nivolumab IV over 30 minutes and ipilimumab IV over 30 minutes on day 1 of each cycle. Cycles repeat every 21 days for 4 cycles. Patients then receive CBM588 PO BID on days 1-28 and nivolumab IV on day 1. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Additionally, patients undergo CT, bone scan and blood sample collection throughout the study. Patients may optionally undergo MRI on study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Scan; Biological: CBM588 Capsules; Procedure: Computed Tomography; Biological: Ipilimumab; Procedure: Magnetic Resonance Imaging; Biological: Nivolumab

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Bone Scan — Undergo bone scan
  Other Names: Bone Scintigraphy
Biological: CBM588 Capsules — Given PO
  Other Names: CBM588; Clostridium butyricum MIYAIRI 588; C. butyricum MIYAIRI 588; C. butyricum strain MIYAIRI 588
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; tomography
Biological: Ipilimumab — Given IV
  Other Names: Anti-Cytotoxic T-Lymphocyte-Associated Antigen-4 Monoclonal Antibody; BMS-734016; Ipilimumab Biosimilar CS1002; MDX-010; MDX-CTLA4; Yervoy
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Biological: Nivolumab — Given IV
  Other Names: ABP 206; BCD-263; BMS-936558; CMAB819; MDX-1106; NIVO; Nivolumab Biosimilar ABP 206; Nivolumab Biosimilar BCD-263; Nivolumab Biosimilar CMAB819; ONO-4538; Opdivo

SUMMARY:
This phase I trial tests the safety, side effects, best dose, and effectiveness of CBM588 in combination with nivolumab and ipilimumab in treating patients with kidney cancer that may have spread from where it first started to nearby tissue, lymph nodes, or distant parts of the body (advanced). CBM588 is a live biotherapeutic that may help improve the effects of immunotherapy. Nivolumab and ipilimumab are monoclonal antibodies that may interfere with the ability of tumor cells to grow and spread by enhancing the ability of the body's immune cells to attack tumor cells. CBM588 in combination with nivolumab and ipilimumab may be safe, tolerable, and/or effective in treating patients with advanced stage kidney cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the safety and tolerability of nivolumab/ipilimumab with escalating doses of Clostridium butyricum MIYAIRI 588 capsules (CBM588) in patients with metastatic renal cell carcinoma.

SECONDARY OBJECTIVES:

I. To evaluate the effect of CBM588 on the clinical efficacy of nivolumab/ipilimumab.

II. To determine the effect of CBM588 (in combination with nivolumab/ipilimumab) in modulation of the gut microbiome in patients with metastatic renal cell carcinoma.

III. To assess the effect of CBM588 on the change of metabolic pathways with the nivolumab/ipilimumab combination in patients with metastatic renal cell carcinoma.

IV. To determine the effect of CBM588 on systemic immunomodulation.

OUTLINE: This is a dose-escalation study of CBM588 followed by a dose-expansion study.

Patients receive CBM588 capsules orally (PO) twice daily (BID) on days 1-21, nivolumab intravenously (IV) over 30 minutes and ipilimumab IV over 30 minutes on day 1 of each cycle. Cycles repeat every 21 days for 4 cycles. Patients then receive CBM588 PO BID on days 1-28 and nivolumab IV on day 1. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Additionally, patients undergo computed tomography (CT), bone scan and blood sample collection throughout the study. Patients may optionally undergo magnetic resonance imaging (MRI) on study.

After completion of study treatment, patients are followed up once a year.

ELIGIBILITY:
Inclusion Criteria:

* Documented informed consent of the participant and/or legally authorized representative

  * Assent, when appropriate, will be obtained per institutional guidelines
* Agreement to allow the use of archival tissue from diagnostic tumor biopsies

  * If unavailable, exceptions may be granted with study principle investigator (PI) approval
* Eastern Cooperative Oncology Group (ECOG) ≤ 2
* Age ≥ 18 years
* Histologically confirmed renal cell carcinoma with clear cell renal cell carcinoma component or sarcomatoid component
* Advanced (not amenable to curative surgery or radiation therapy) or metastatic (American Joint Committee on Cancer [AJCC] stage IV) renal cell carcinoma with intermediate- or poor-risk disease by International Metastatic Renal Cell Carcinoma Database Consortium (IMDC) criteria
* No prior systemic therapy for renal cell carcinoma (RCC) with the following exception:

  * One prior adjuvant or neoadjuvant therapy for completely resectable RCC if recurrence occurred at least 6 months after the last dose of adjuvant or neoadjuvant therapy
* Measurable disease by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1
* Fully recovered from the acute toxic effects (except alopecia) to ≤ grade 1 to prior anti-cancer therapy
* Absolute neutrophil count (ANC) ≥ 1500/uL without granulocyte colony-stimulating factor support
* White blood cell count ≥ 2500/uL
* Platelets ≥ 100,000/uL without transfusion
* Hemoglobin ≥ 8 g/dL
* Alanine aminotransferase (ALT), aspartate aminotransferase (AST), and alkaline phosphatase (ALP) ≤ 3 x upper limit of normal (ULN). ALP ≤ 5 x ULN with documented bone metastases
* Total bilirubin ≤ 1.5 x ULN (for subjects with Gilbert's disease ≤ 3 x ULN)
* Serum albumin ≥ 2.8 g/dl
* Prothrombin time (PT)/international normalized ratio (INR) or partial thromboplastin time (PTT) test < 1.3 x the laboratory ULN
* Serum calculated creatinine clearance ≥ 50mL/min using the Cockcroft-Gault equation
* Sexually active fertile subjects and their partners must agree to use medically accepted methods of contraception (e.g., barrier methods, including male condom, female condom, or diaphragm with spermicidal gel) during the course of the study and for 5 months after the last dose of nivolumab for women with childbearing potential, and 7 months after the last dose of nivolumab for men
* Female subjects of childbearing potential must not be pregnant at screening. Female subjects are considered to be of childbearing potential unless one of the following criteria is met: documented permanent sterilization (hysterectomy, bilateral salpingectomy, or bilateral oophorectomy) or documented postmenopausal status (defined as 12 months of amenorrhea in a woman > 45 years-of-age in the absence of other biological or physiological causes. In addition, females < 55 years-of-age must have a serum follicle stimulating (FSH) level > 40 mIU/mL to confirm menopause).

  * Note: Documentation may include review of medical records, medical examinations, or medical history interview by study site

Exclusion Criteria:

* Prior treatment with ipilimumab and/or nivolumab
* Current use, or intent to use, probiotics, yogurt, or bacterial fortified foods during the period of treatment
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to study agent
* Active interstitial lung disease (ILD)/pneumonitis or history of ILD/pneumonitis requiring treatment with systemic steroids
* Known medical condition (e.g., a condition associated with diarrhea or acute diverticulitis) that, in the investigator's opinion, would increase the risk associated with study participation or study drug administration or interfere with the interpretation of safety results
* Receipt of any type of cytotoxic, biologic, or other systemic anticancer therapy (including investigational) within 4 weeks before first dose of study treatment
* Radiation therapy for bone metastasis within 2 weeks or any other radiation therapy within 4 weeks before first dose of study treatment. Systemic treatment with radionuclides within 6 weeks before first dose of study treatment. Subjects with clinically relevant ongoing complications from prior radiation therapy are not eligible
* Known brain metastases or cranial epidural disease unless adequately treated with radiotherapy and/or surgery (including radiosurgery) and stable for at least 4 weeks prior to first dose of study treatment after radiotherapy or at least 4 weeks prior to first dose of study treatment after major surgery (e.g., removal or biopsy of brain metastasis). Subjects must have complete wound healing from major surgery or minor surgery before first dose of study treatment. Eligible subjects must be neurologically asymptomatic and without corticosteroid treatment at the time of first dose of study treatment
* Administration of a live, attenuated vaccine within 30 days before first dose of study treatment
* The subject has uncontrolled, significant intercurrent or recent illness including, but not limited to, the following conditions:

  * Any condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalent) or other immunosuppressive medications within 14 days before first dose of study treatment. Note: Inhaled, intranasal, intra-articular, or topical steroids are permitted. Adrenal replacement steroid doses ≤ 10 mg daily prednisone equivalent are permitted. Transient short-term use of systemic corticosteroids for allergic conditions (e.g., contrast allergy) is also allowed
  * Active infection requiring systemic treatment. Acute or chronic hepatitis B or C infection, known human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS)-related illness requiring systemic treatments, or known positive test for tuberculosis infection where there is clinical or radiographic evidence of active mycobacterial infection
  * History of idiopathic pulmonary fibrosis, organizing pneumonia, drug-induced pneumonitis, idiopathic pneumonitis, or evidence of active pneumonitis on screening chest CT scan
  * Malabsorption syndrome
  * Uncompensated/symptomatic hypothyroidism
  * Moderate to severe hepatic impairment (Child-Pugh B or C)
  * Requirement for hemodialysis or peritoneal dialysis
  * History of solid organ or allogenic stem cell transplant
  * Other clinically significant disorders that would preclude safe study participation

    * Any active, known, or suspected autoimmune disease will be excluded, with the following exceptions:

      * Type 1 diabetes mellitus
      * Hypothyroidism only requiring hormone replacement
      * Skin disorders (e.g., vitiligo, psoriasis, or alopecia) not requiring systemic treatment
      * Conditions not expected to recur in the absence of an external trigger
* Pregnant or lactating females
* Inability to swallow tablets/capsules or unwillingness or inability to receive IV administration
* Previously identified allergy or hypersensitivity to components of the study treatment formulations or history of severe infusion-related reactions to monoclonal antibodies. Subjects with rare hereditary problems of galactose intolerance, the Lapp lactase deficiency or glucose-galactose malabsorption are also excluded
* Any other active malignancy at time of first dose of study treatment or diagnosis of another malignancy within 3 years prior to first dose of study treatment that requires active treatment, except for locally curable cancers that have been apparently cured, such as basal or squamous cell skin cancer, superficial bladder cancer, or carcinoma in situ of the prostate, cervix, or breast
* Exclusion of subjects with a history of myocarditis or congestive heart failure (as defined by New York Heart Association Functional Classification III or IV), as well as unstable angina, serious uncontrolled cardiac arrhythmia, uncontrolled infection, or myocardial infarction 6 months prior to study entry
* Exclusion of subjects whose baseline pulse oximetry is less than 92% on room air
* Any other condition that would, in the investigator's judgment, contraindicate the patient's participation in the clinical study due to safety concerns with clinical study procedures
* Prospective participants who, in the opinion of the investigator, may not be able to comply with all study procedures (including compliance issues related to feasibility/logistics)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2024-06-19 (Estimated); Primary Completion 2026-10-19 (Estimated); Study Completion 2026-10-19 (Estimated)

PRIMARY OUTCOMES:
Dose limiting toxicity (DLT) | Up to 28 days
  Toxicities at least possibly related to study agent will be graded according to National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) version (v)5.0.
Maximum tolerated dose (MTD) | Up to 28 days
  MTD estimate will be the highest dose with the occurrence of DLT in no more than 1 out of 6 of the patients.
Incidence of adverse events (AEs) | Up to 3 years
  AEs will be graded using CTCAE. Summaries will be provided overall and by dose group. The number and percentage of subjects reporting treatment-emergent AEs (TEAE) will be summarized overall and by the worse CTCAE grade, with a breakdown by dose. The number and percentage of subjects reporting TEAEs considered related to each study drug will be summarized.

SECONDARY OUTCOMES:
Progression free survival (PFS) | From enrollment to progression or death, assessed up to 3 years
  PFS will be defined as the duration of time from start of treatment to time of progressive disease or death, whichever occurs first. PFS will be estimated using the Kaplan-Meier method. The difference in PFS across dose levels will be explored using the log-rank test. Median PFS time for each dose level will be reported, and the Cox proportional hazard model will be used to estimate the hazard ratio and its confidence interval without adjustment for clinically relevant covariates.
Overall response rate (ORR) | Up to 3 years
  Evaluated using Response Evaluation Criteria in Solid Tumors (RECIST) v1.1. The best overall response is the best response recorded from the start of the treatment until disease progression or recurrence. ORR will be calculated as the number of patients with complete or partial response divided by the total number of treated/evaluable subjects. ORR will be summarized by dose levels, number, and percentage, along with corresponding exact 95% confidence interval. The association between dose level and overall response as per RECIST v1.1 criteria will be examined using Fisher's exact test.
Change in stool microbial diversity | Baseline to week 12 of therapy
  The Shannon index will be computed from whole metagenome sequence data from stool samples to compare microbial diversity between baseline and 12 weeks and between the two study arms. The index takes into account the number of species (richness) and their relative abundance (evenness). A higher Shannon index indicates greater microbial diversity. The minimum value the Shannon diversity index can take is 0 (one species) and there is no upper limit to the index.
Change in abundancies of gut microbiome species | Baseline to week 12 of therapy
  The taxonomic composition of the microbiome will be determined from whole metagenome sequencing of stool samples and the relative abundancies of species will be compared between baseline and 12 weeks and between the two study arms. The relative abundancies will vary from 0 to 1.
Metabolic pathways | Baseline to week 12 of therapy
  The abundancies of gut microbiome metabolic pathways will be estimated using whole metagenome sequence data from stool samples. Metabolic pathways with significantly different counts between baseline and week 12 and between the two study arms will be compared.
Changes in serum short chain fatty acids | Baseline up to 3 years of therapy
  The proportion of serum short chain fatty acids will be estimated using translational methods. The levels (ng/ml) of butyrate and other short chain fatty acids in blood will be assessed graphically over serial timepoints of blood collection to determine trends over time and between study arms.
Circulating regulatory T cells (Tregs) and myeloid-derived suppressor cells (MDSCs) | Baseline up to 3 years of therapy
  The proportion of Tregs and MDSCs in the blood will be estimated using flow cytometry methods. The percentage of viable immune cells (from 0%-100%) will be assessed graphically over serial timepoints of blood collection to determine trends over time and between study arms.
Serum Cytokines | Baseline up to 3 years of therapy
  The levels (pg/ml) of serum cytokines in blood will be estimated using flow cytometry methods and will include IFN gamma, TNF alpha, IL-2, IL-6, IL-8, IL-10, GM-CSF, and other cytokines/chemokines. The relative levels of cytokines will be assessed graphically over serial timepoints of blood collection to determine trends over time and between study arms.

CONTACTS AND LOCATIONS:
Overall Officials: Alex Chehrazi-Raffle, MD, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States

REFERENCES:
- [Background] Dizman N, Meza L, Bergerot P, Alcantara M, Dorff T, Lyou Y, Frankel P, Cui Y, Mira V, Llamas M, Hsu J, Zengin Z, Salgia N, Salgia S, Malhotra J, Chawla N, Chehrazi-Raffle A, Muddasani R, Gillece J, Reining L, Trent J, Takahashi M, Oka K, Higashi S, Kortylewski M, Highlander SK, Pal SK. Nivolumab plus ipilimumab with or without live bacterial supplementation in metastatic renal cell carcinoma: a randomized phase 1 trial. Nat Med. 2022 Apr;28(4):704-712. doi: 10.1038/s41591-022-01694-6. Epub 2022 Feb 28. PMID 35228755
- [Background] Tomita Y, Ikeda T, Sakata S, Saruwatari K, Sato R, Iyama S, Jodai T, Akaike K, Ishizuka S, Saeki S, Sakagami T. Association of Probiotic Clostridium butyricum Therapy with Survival and Response to Immune Checkpoint Blockade in Patients with Lung Cancer. Cancer Immunol Res. 2020 Oct;8(10):1236-1242. doi: 10.1158/2326-6066.CIR-20-0051. Epub 2020 Jul 14. PMID 32665261
- [Background] Tomita Y, Goto Y, Sakata S, Imamura K, Minemura A, Oka K, Hayashi A, Jodai T, Akaike K, Anai M, Hamada S, Iyama S, Saruwatari K, Saeki S, Takahashi M, Ikeda T, Sakagami T. Clostridium butyricum therapy restores the decreased efficacy of immune checkpoint blockade in lung cancer patients receiving proton pump inhibitors. Oncoimmunology. 2022 May 27;11(1):2081010. doi: 10.1080/2162402X.2022.2081010. eCollection 2022. PMID 35655708
- [Background] Tomita Y, Sakata S, Imamura K, Iyama S, Jodai T, Saruwatari K, Hamada S, Akaike K, Anai M, Fukusima K, Takaki A, Tsukamoto H, Goto Y, Motozono C, Sugata K, Satou Y, Ueno T, Ikeda T, Sakagami T. Association of Clostridium butyricum Therapy Using the Live Bacterial Product CBM588 with the Survival of Patients with Lung Cancer Receiving Chemoimmunotherapy Combinations. Cancers (Basel). 2023 Dec 21;16(1):47. doi: 10.3390/cancers16010047. PMID 38201474
- [Background] Paz Del Socorro T, Oka K, Boulard O, Takahashi M, Poulin LF, Hayashi A, Chamaillard M. The biotherapeutic Clostridium butyricum MIYAIRI 588 strain potentiates enterotropism of Rorgammat+Treg and PD-1 blockade efficacy. Gut Microbes. 2024 Jan-Dec;16(1):2315631. doi: 10.1080/19490976.2024.2315631. Epub 2024 Feb 22. PMID 38385162